CLINICAL TRIAL: NCT01818934
Title: Ultrasound Screening for Developmental Dysplasia of the Hip in the Neonate: The Effect on Treatment Rate and Prevalence of Late Cases
Brief Title: Ultrasound Screening for Developmental Dysplasia of the Hip in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Institute of Child Health (Other)
Responsible Party: Principal Investigator, Lene Bjerke Laborie, MD, Phd, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 3.2006.144
Record Dates: First submitted 2013-03-21; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Hip Dysplasia
Keywords: hip dysplasia; screening
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- expert clinical exam only (Active Comparator): all babies assigned to this group had expert clinical examination only, no hip ultrasound
  Interventions: Procedure: hip ultrasound
- selective hip ultrasound screening (Active Comparator): all children classified at increased risk, based on clinical findings and/or risk factors (breech presentation, family history, foot deformity)received a hip ultrasound at birth, in addition to expert clinical screening
  Interventions: Procedure: hip ultrasound
- universal hip ultrasound screening (Active Comparator): All newborns assigned to this arm received hip ultrasound at birth in addition to expert clinical examination
  Interventions: Procedure: hip ultrasound

INTERVENTIONS:
Procedure: hip ultrasound — Standardized single-examiner Hip ultrasound was offered to all babies in the universal group, babies at increased risk in the selective group, and to no babies in the clinical exam only group

SUMMARY:
The aim of the randomized controlled trial was to determine whether the addition of a general or of a selective ultrasound screening program resulted in more appropriate criteria for treatment and a reduced prevalence of late DDH compared with clinical examination alone.

DETAILED DESCRIPTION:
This is a retrospective registration of a RCT carried out in 1988-90, with a IRB approved follow-up at skeletal maturity carried out in 2007-09. Both the RCT and the follow-up study were carried out in the same institution, by the same PI (Prof. Karen Rosendahl) and her co-workers.

Detailed information is published in the following paper:

Rosendahl K, Markestad T, Lie RT. Ultrasound screening for developmental dysplasia of the hip in the neonate: the effect on treatment rate and prevalence of late cases. Pediatrics 1994;94:47-52.

A sample of the initial RCT was invited for a maturity review/follow-up at skeletal maturity.

The follow-up at skeletal maturity is called:

Radiological indices of hip dysplasia and osteoarthritis at skeletal maturity in the Bergen Birth Cohort. Associations with neonatal hip dysplasia, childhood growth and genetic predisposition

and is included in the approval by the Regional Ethical Committee for Medical and Health Research (No 3.2006.144). All participants of the follow-up study gave written informed consent according to the 1964 Declaration of Helsinki.

The follow-up had the following main aims:

1) estimate the prevalence of radiologically defined hip dysplasia, femoroacetabular impingement and osteoarthritis assessed at skeletal maturity 2)report the frequency of 4 longitudinal dysplasia phenotypes based on sonographic assessments in the newborn and radiological assessments at skeletal maturity 3)investigate associations of dysplasia as defined in 1 and 2 above in univariate and multivariate models with clinically assessed hip joint mobility/joint hypermobility, weight, height and body mass index (BMI) at age 18/19 years, prepubertal weight, height and BMI trajectories using data from child health records, first degree family history of hip dysplasia with or without hip arthroplasty, perinatal factors, measures of OA including minimum joint space, acetabular depth ratio and reported hip pain 5) establish a genetic resource by obtaining and archiving salivary DNA samples.

ELIGIBILITY:
Inclusion Criteria:

* all babies born at our institution during 1/1988-06/1990

Exclusion Criteria:

* low birthweight <1500 grams, severe malformations, death within first month

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11925 (Actual)
Dates: Start 1988-01; Primary Completion 1990-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
prevalence of DDH detected after newborn period | 20 years
  prevalence of late cases of DDH, detected after newborn period (after first month of age, including in childhood as assessed in original RCT during 1988-90, with a minimum follow-up time of 27 months, and also at skeletal maturity, as assessed in follow-up study during 2007-09.

SECONDARY OUTCOMES:
treatment rate | 20 years
  abduction treatment and/or surgery during infancy, later childhood and skeletal maturity

OTHER OUTCOMES:
avascular necrosis of femoral head (AVN) | 20 years
  avascular necrosis of femoral head (AVN) as a complication to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Rosendahl, Prof, Principal Investigator — Pediatric section, Department of Radiology, Haukeland University hospital, University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Bergen, Norway

REFERENCES:
- [Result] Rosendahl K, Markestad T, Lie RT. Ultrasound screening for developmental dysplasia of the hip in the neonate: the effect on treatment rate and prevalence of late cases. Pediatrics. 1994 Jul;94(1):47-52. PMID 8008537
- [Result] Laborie LB, Engesaeter IO, Lehmann TG, Sera F, Dezateux C, Engesaeter LB, Rosendahl K. Radiographic measurements of hip dysplasia at skeletal maturity--new reference intervals based on 2,038 19-year-old Norwegians. Skeletal Radiol. 2013 Jul;42(7):925-35. doi: 10.1007/s00256-013-1574-y. Epub 2013 Jan 27. PMID 23354528
- [Result] Laborie LB, Lehmann TG, Engesaeter IO, Eastwood DM, Engesaeter LB, Rosendahl K. Prevalence of radiographic findings thought to be associated with femoroacetabular impingement in a population-based cohort of 2081 healthy young adults. Radiology. 2011 Aug;260(2):494-502. doi: 10.1148/radiol.11102354. Epub 2011 May 25. PMID 21613440
- [Result] Laborie LB, Lehmann TG, Engesaeter IO, Engesaeter LB, Rosendahl K. Is a positive femoroacetabular impingement test a common finding in healthy young adults? Clin Orthop Relat Res. 2013 Jul;471(7):2267-77. doi: 10.1007/s11999-013-2850-9. Epub 2013 Feb 15. PMID 23412733
- [Result] Engesaeter IO, Laborie LB, Lehmann TG, Sera F, Fevang J, Pedersen D, Morcuende J, Lie SA, Engesaeter LB, Rosendahl K. Radiological findings for hip dysplasia at skeletal maturity. Validation of digital and manual measurement techniques. Skeletal Radiol. 2012 Jul;41(7):775-85. doi: 10.1007/s00256-011-1283-3. Epub 2011 Sep 25. PMID 21946945
- [Result] Engesaeter IO, Laborie LB, Lehmann TG, Fevang JM, Lie SA, Engesaeter LB, Rosendahl K. Prevalence of radiographic findings associated with hip dysplasia in a population-based cohort of 2081 19-year-old Norwegians. Bone Joint J. 2013 Feb;95-B(2):279-85. doi: 10.1302/0301-620X.95B2.30744. PMID 23365042
- [Derived] Laborie LB, Engesaeter IO, Lehmann TG, Eastwood DM, Engesaeter LB, Rosendahl K. Screening strategies for hip dysplasia: long-term outcome of a randomized controlled trial. Pediatrics. 2013 Sep;132(3):492-501. doi: 10.1542/peds.2013-0911. Epub 2013 Aug 19. PMID 23958776